CLINICAL TRIAL: NCT03075319
Title: Use of Perioperative Photograph as a Motivation for Increasing Range of Motion After Primary Total Knee Arthroplasty: Randomized Controlled Trial
Brief Title: Use of Perioperative Photograph as a Motivation for Increasing Range of Motion After Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Boontanapibul, Krit, M.D. (Individual)
Responsible Party: Principal Investigator, piya pinsornsak, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-OT-6-049/56
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received perioperative photograph (Experimental): Perioperative knee range of motion (ROM) were measured with long arm goniometer immediately after close the wound. Perioperative knee photographs in full flexion and extension positions were taken and gave to experimental group in the day after surgery.
  Interventions: Procedure: Received perioperative photograph
- Didn't receive perioperative photograph (Active Comparator): Perioperative knee range of motion (ROM) were measured with long arm goniometer immediately after close the wound. Perioperative knee photographs in full flexion and extension positions were taken but participants in this group didn't receive perioperative photographs.
  Interventions: Procedure: Didn't receive perioperative photograph

INTERVENTIONS:
Procedure: Received perioperative photograph — All participants in experimental group were adviced to see periopertive knee photograph before rehabilitation everyday.
  Postoperative knee ROM were recorded at day 3, 6 week, 3 month and 6 month. Flexion and extension angle were measured with long arm goniometer.
  The outcome assessors were blinded to treatment groups.
  Arms: Received perioperative photograph
Procedure: Didn't receive perioperative photograph — All participants in active comparator group didn't receive perioperative knee photograph.
  Postoperative knee ROM were recorded at day 3, 6 week, 3 month and 6 month. Flexion and extension angle were measured with long arm goniometer.
  The outcome assessors were blinded to treatment groups.
  Arms: Didn't receive perioperative photograph

SUMMARY:
Total knee arthroplasty (TKA) is recognized as a successful procedure for treating osteoarthritis (OA) of the knee. One important factor that make the successful surgery is the degree of knee flexion. Providing more range of motion after TKA impact on the convenience of daily of life such as climbing stairs, sitting on the floor particularly in Asian cultures which require a lot of ground activities. Data are limited on the added benefits of perioperative photograph as motivation for increasing range of motion after TKA.

Half of participants received perioperative photograph as motivation, while the other half did not after total knee arthroplasty.

DETAILED DESCRIPTION:
All participants received spinal anesthesia, multimodal local anesthetic infiltration and patient controlled analgesia (PCA) for 24 hours post surgery. The surgical techniques, postoperative medications and rehabilitation protocols were identical in both groups. Perioperative knee range of motion (ROM) were measured with long arm goniometer immediately after close the wound. Perioperative knee photographs in full flexion and extension positions were taken and were given to experimental group in the day after surgery. Postoperative knee ROM were recorded at day 3, 6 week, 3 month and 6 month. The outcome assessors were blinded to treatment groups during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Primary OA of the knee, aged less than 80 years old, and able to understand and comply with the study procedures.

Exclusion Criteria:

* Knee range of motion less than 90 degrees
* Psychotic disorders
* History of stroke
* Inability to undergo a spinal block

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Knee range of motion | Flexion and extension angle at 6 month
  Compare flexion and extension angle using long arm goniometer between experimental and active comparator group

SECONDARY OUTCOMES:
Knee society scores | 6 week, 3 month and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Piya Pinsornsak, Principal Investigator — Faculty of Medicine, Thammasat university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ritter MA, Campbell ED. Effect of range of motion on the success of a total knee arthroplasty. J Arthroplasty. 1987;2(2):95-7. doi: 10.1016/s0883-5403(87)80015-3. PMID 3612145
- [Result] Miner AL, Lingard EA, Wright EA, Sledge CB, Katz JN; Kinemax Outcomes Group. Knee range of motion after total knee arthroplasty: how important is this as an outcome measure? J Arthroplasty. 2003 Apr;18(3):286-94. doi: 10.1054/arth.2003.50046. PMID 12728419
- [Result] Meneghini RM, Pierson JL, Bagsby D, Ziemba-Davis M, Berend ME, Ritter MA. Is there a functional benefit to obtaining high flexion after total knee arthroplasty? J Arthroplasty. 2007 Sep;22(6 Suppl 2):43-6. doi: 10.1016/j.arth.2007.03.011. Epub 2007 Jul 26. PMID 17823014
- [Result] Kurosaka M, Yoshiya S, Mizuno K, Yamamoto T. Maximizing flexion after total knee arthroplasty: the need and the pitfalls. J Arthroplasty. 2002 Jun;17(4 Suppl 1):59-62. doi: 10.1054/arth.2002.32688. PMID 12068407
- [Result] Fisher DA, Dierckman B, Watts MR, Davis K. Looks good but feels bad: factors that contribute to poor results after total knee arthroplasty. J Arthroplasty. 2007 Sep;22(6 Suppl 2):39-42. doi: 10.1016/j.arth.2007.04.011. Epub 2007 Jul 26. PMID 17823013
- [Result] Harvey IA, Barry K, Kirby SP, Johnson R, Elloy MA. Factors affecting the range of movement of total knee arthroplasty. J Bone Joint Surg Br. 1993 Nov;75(6):950-5. doi: 10.1302/0301-620X.75B6.8245090.
- [Result] Ritter MA, Harty LD, Davis KE, Meding JB, Berend ME. Predicting range of motion after total knee arthroplasty. Clustering, log-linear regression, and regression tree analysis. J Bone Joint Surg Am. 2003 Jul;85(7):1278-85. doi: 10.2106/00004623-200307000-00014. PMID 12851353
- [Result] Dennis DA, Komistek RD, Stiehl JB, Walker SA, Dennis KN. Range of motion after total knee arthroplasty: the effect of implant design and weight-bearing conditions. J Arthroplasty. 1998 Oct;13(7):748-52. doi: 10.1016/s0883-5403(98)90025-0. PMID 9802659
- [Result] Sharma L, Sinacore J, Daugherty C, Kuesis DT, Stulberg SD, Lewis M, Baumann G, Chang RW. Prognostic factors for functional outcome of total knee replacement: a prospective study. J Gerontol A Biol Sci Med Sci. 1996 Jul;51(4):M152-7. doi: 10.1093/gerona/51a.4.m152. PMID 8680997
- [Result] Bonnin M, Laurent JR, Parratte S, Zadegan F, Badet R, Bissery A. Can patients really do sport after TKA? Knee Surg Sports Traumatol Arthrosc. 2010 Jul;18(7):853-62. doi: 10.1007/s00167-009-1009-4. Epub 2009 Dec 24. PMID 20033676
- [Result] Naylor JM, Ko V, Adie S, Gaskin C, Walker R, Harris IA, Mittal R. Validity and reliability of using photography for measuring knee range of motion: a methodological study. BMC Musculoskelet Disord. 2011 Apr 18;12:77. doi: 10.1186/1471-2474-12-77. PMID 21496347
- [Result] Gogia PP, Braatz JH, Rose SJ, Norton BJ. Reliability and validity of goniometric measurements at the knee. Phys Ther. 1987 Feb;67(2):192-5. doi: 10.1093/ptj/67.2.192. PMID 3809242